CLINICAL TRIAL: NCT00893477
Title: An Open Label, Multicenter, Non Randomized Phase II Study to Evaluate Anti-tumor Efficacy and Safety of GM-CSF (Sargramostim, Leukine®) Associated With Rituximab (MabThera®) in Patients With Follicular Non Hodgkin's Lymphoma With no Prior Treatment
Brief Title: GM-CSF and Rituximab in Treating Patients With Previously Untreated Follicular Non-Hodgkin Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: French Innovative Leukemia Organisation (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: GOELAMS-FL2008-RGM; CDR0000637112 (Registry Identifier: PDQ (Physician Data Query)); EUDRACT-2007-005580-95; RECF0906
Record Dates: First submitted 2009-05-05; First posted 2009-05-06 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2009-07

CONDITIONS: Lymphoma
Keywords: stage II grade 1 follicular lymphoma; stage II grade 2 follicular lymphoma; stage II grade 3 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — Rituximab; sargramostim; Gene Expression Profiling; Gene Rearrangement; Polymerase Chain Reaction; Amplified Fragment Length Polymorphism Analysis

INTERVENTIONS:
Biological: rituximab
Biological: sargramostim
Genetic: gene expression analysis
Genetic: gene rearrangement analysis
Genetic: polymerase chain reaction
Genetic: polymorphism analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Biological therapies, such as GM-CSF, may stimulate the immune system in different ways and stop cancer cells from growing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving GM-CSF together with rituximab may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving GM-CSF together with rituximab works in treating patients with previously untreated follicular non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the clinical efficacy of sargramostim (GM-CSF) and rituximab, in terms of overall objective complete and partial response rates, in patients with previously untreated follicular non-Hodgkin lymphoma.

Secondary

* Evaluate the time to progression in patients treated with this regimen.
* Evaluate the overall survival of patients treated with this regimen.
* Evaluate the duration of response in patients treated with this regimen.
* Evaluate the safety profile of this regimen in these patients.
* Evaluate the influence of FcγR polymorphisms on clinical response.
* Monitor FcγR-expressing cells in peripheral blood during treatment.
* Monitor the molecular biological marker bcl2 [t(14;18)] in peripheral blood and bone marrow.

OUTLINE: This is a multicenter study.

* Induction therapy: Patients receive sargramostim (GM-CSF) subcutaneously (SC) on days 1-5 and rituximab IV on day 1. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.
* Maintenance therapy: Patients receive GM-CSF SC on days 1-5 and rituximab IV on day 1. Treatment repeats every 8 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.

Blood and bone marrow samples are collected at baseline and periodically during study for analysis of bcl2 rearrangement by PCR assay; FcγR expression by immunophenotyping; and FcγR polymorphisms.

After completion of study therapy, patients are followed every 3 months for 1 year and then every 6 months for up to 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically and immunophenotypically confirmed CD20+ follicular lymphoma according to WHO classification

  * Grade 1-3a disease
  * Stage II-IV disease
  * Non-bulky disease
* Must have undergone initial nodal biopsy within the past 4 months
* At least 1 measurable lesion
* Low tumor-burden, as defined by the following GELF criteria:

  * Nodal or extranodal tumor mass (diameter < 7 cm)
  * No systemic B symptoms
  * No increased LDH and β2 microglobulinemia
  * No substantial splenic enlargement
  * No serous effusion
  * No compression syndrome

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active hepatitis

PRIOR CONCURRENT THERAPY:

* No prior treatment, including steroids and radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-03; Primary Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Overall objective tumor response rate at the end of induction therapy

SECONDARY OUTCOMES:
Time to progression
Overall survival
Duration of response
Time to next treatment
Safety profile
Influence of FcγR polymorphisms on clinical response and survival
FcγR expression during study treatment
Molecular biological marker bcl2 [t(14;18)] in peripheral blood and bone marrow as measured by PCR assay

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Francois Rossi, MD, PhD, Principal Investigator — Hopital Lapeyronie-CHU Montpellier